CLINICAL TRIAL: NCT04325516
Title: Decoding Motion Planning Using Cortical Potentials in People With a Transfemoral Amputation and Able-bodied Individuals
Brief Title: Decoding Motion Planning Using Cortical Potentials
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Jo Ghillebert, Principle Investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EEGstudy
Record Dates: First submitted 2020-03-20; First posted 2020-03-27 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Lower Limb Amputation Above Knee (Injury)
Keywords: Amputee; Lower limb; Brain activity; Cortical potentials; Movement intention
MeSH Terms: conditions — Wounds and Injuries | interventions — Activities of Daily Living

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People with a lower limb amputation (Experimental): Participants will perform four tasks in a randomized order:
  * sit to stand
  * dorsi flexion of the foot
  * knee extension
  * hip extension
  Interventions: Behavioral: Daily activities
- Able bodied individuals (Experimental): Participants will perform four tasks in a randomized order:
  * sit to stand
  * dorsi flexion of the foot
  * knee extension
  * hip extension
  Interventions: Behavioral: Daily activities

INTERVENTIONS:
Behavioral: Daily activities — Participants will perform four tasks in a randomized order:
  * sit to stand
  * dorsi flexion of the foot
  * knee extension
  * hip extension

SUMMARY:
The team will investigate the user's intention to move by using cortical activity during a sit to stand movement performance in people with a transfemoral amputation and able-bodied individuals. The goal is to get insights in pre-movement onset indicators within the brain that initiate the sit to stand transfer. The hypothesis is that people with a transfemoral amputation use different brain locations for motion planning compared to able-bodied individuals.

DETAILED DESCRIPTION:
The evolution of lower limb prostheses has made considerable progress in the past decades. There has been a transition from passive (e.g. Total knee®, Össur) to quasi-passive (e.g. C-leg®, Otto Bock) and eventually to active prostheses (e.g. Power knee®, Össur). The development always focused on an amputation as a primary peripheral disorder. For example, manufacturers have been searching to compensate the loss of muscle mass by adding torque into the prosthesis. However, few considerations have yet been taken to the fact that central adaptations are also observed after amputation in terms of neuroplasticity and reorganization.

The atypical motion planning strategies of people with a lower limb amputation (LLA) could possibly be related to the challenges that they experience during daily activities, such as the sit to stand transfer. Standing up from a chair is a relevant clinical problem and current devices do not yet relieve the asymmetrical loading. A few studies have already investigated the muscular activity during a sit to stand movement in people with a LLA and able-bodied individuals. The movement is characterized by a forward displacement of the centre of mass with the highest activation of the m. gluteus maximus, m. adductor magnus and m. biceps femoris.The sit to stand transfer is a potential movement to investigate brain activity incorporating the advantages and disadvantages of EEG measurements.

Until now, the development of lower limb prostheses approaches people with a LLA as a peripheral disorder whereas relevant central adaptations are also observed. Therefore, the purpose of this study is to identify the cortical activity that is responsible for successfully completing a sit to stand transfer. The hypothesis is that different brain locations are activated in people with a transfemoral amputation for motion planning compared to able-bodied individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25 - 75 years
* Gender: men and women
* Level of amputation: unilateral transfemoral
* Vascular or traumatic cause of amputation
* Medicare Functional Classification Level25: K3-4
* Participants are able to stand up from a chair and return to the seated position without support of their hands for ten repetitions
* Participants wear their prosthesis for at least 8 hours/day (Prosthetic use has been shown to have an influence on functional reorganization)
* No cognitive impairment. This will be objectified with the mini-mental state examination (score on 30)

Exclusion Criteria:

* Any neurological disease
* No upper limb or bilateral amputation

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
ElectroEncephalography in milliseconds | Approximatley 9 months
  Movement related cortical potential before the actual movement
ElectroMyography activity in milliseconds | Approximatley 9 months
  Amplitude
ElectroMyography timing | Approximatley 9 months
  Time of movement onset

SECONDARY OUTCOMES:
Duration of the sit to stand test | Approximatley 9 months
  Duration of the sit to stand test

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No